CLINICAL TRIAL: NCT04789122
Title: Assessment of Poles' Attitudes Towards Living Kidney Donation
Status: Completed | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Paulina Kurleto, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: WLNZ/NoZ/4/2020
Record Dates: First submitted 2021-02-26; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Attitude assessment — The study covered a representative group of 1000 people. Own questionnaire and standardized tools sent online via the Statistical Research and Analysis Office, in compliance with the privacy policy and personal data protection of the General Data Protection Regulation.

SUMMARY:
The main goal of the project is to examine the public opinion on living kidney donation and to assess the knowledge of Poles in this field.

DETAILED DESCRIPTION:
Researchers also want to estimate how large percentage of the respondents will declare their willingness to donate a kidney to a stranger and what percentage of respondents would support a possible extension of the existing law on the collection, storage and transplantation of cells, tissues and organs of July 1, 2005 to include donation to a stranger.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Polish citizenship

Exclusion Criteria:

* below 18 yers of age
* not Polish citizen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Poles randomly chosen from all voivodships,
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Questionnaire answers under statistical processing | 15.03.2021

CONTACTS AND LOCATIONS:
Locations (1):
- Andrzej Frycz Modrzewski Krakow University, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kurleto P, Tomaszek L, Milaniak I, Bramstedt KA. Polish attitudes towards unspecified kidney donation: a cross-sectional study. BMC Nephrol. 2022 Apr 13;23(1):142. doi: 10.1186/s12882-022-02767-x. PMID 35418039
- [Derived] Kurleto P, Tomaszek L, Milaniak I, Medrzycka-Dabrowska W. Factors Associated with the Willingness to Become a Living Kidney Donor: A National Cross-Sectional Study. Int J Environ Res Public Health. 2022 Jan 25;19(3):1313. doi: 10.3390/ijerph19031313. PMID 35162337